CLINICAL TRIAL: NCT02321670
Title: Scandinavian Urethroplasty Study. A Multicentre, Prospective, Randomized Study Comparing Bulbar Urethroplasty With Excision and Primary Anastomosis or With an Onlay Grafting Procedure Using Buccal Mucosa.
Brief Title: Scandinavian Urethroplasty Study
Acronym: SUPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sahlgrenska University Hospital (Other); Region Örebro County (Other); Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Ole Jacob Nilsen, Consultant, Head of section, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OUS-URO-SUPS
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Urethral Stricture
Keywords: operative technique
MeSH Terms: conditions — Urethral Stricture | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- End-to-end (Active Comparator): Excision of the stricture and end-to-end anastomosis of the urethra.
  Interventions: Procedure: End-to-end
- Graft (Active Comparator): Incision of the stricture and grafting procedure with buccal mucosa where the corpus spongiosum is not divided.
  Interventions: Procedure: Graft

INTERVENTIONS:
Procedure: End-to-end — Excision of the stricture and end-to-end anastomosis of the urethra.
  Arms: End-to-end
Procedure: Graft — Incision of stricture and grafting procedure with buccal mucosa where the corpus spongiosum is not divided
  Arms: Graft

SUMMARY:
A multicentre, prospective, randomized study comparing bulbar urethroplasty with excision and primary anastomosis or with an onlay grafting procedure using buccal mucosa.

DETAILED DESCRIPTION:
The study is a prospective, randomized study to compare two common techniques of urethroplasty used to treat bulbar urethral strictures. One technique is excision of the stricture and end-to-end anastomosis of the urethra. The other technique is an onlay grafting procedure with buccal mucosa where the corpus spongiosum is not divided. The study is designed to compare complications of sexual and penile function, and is not powered to compare the success rates of the two techniques. The primary endpoint will be degree of erectile dysfunction and penile complications. The secondary endpoint will be restricturing leading to reoperation, and other complications.

ELIGIBILITY:
Inclusion Criteria:

Patient with bulbar urethral stricture, length estimated by urethrography or endoscopy ≤ 2 cm

Patient is able and willing to sign informed consent

Patient is able and willing to complete all study requirements

Exclusion Criteria:

Previous open urethroplasty

Previous hypospadia surgery

Previous surgery for congenital curvature or Mb Peyronie

Previous pelvic irradiation therapy

Known grave psychiatric disorder

Haemophilia or other clotting disorders that cause bleeding diathesis

Use of medication to increase erectile function, such as PDE5-inhibitors and intracavernous injections, during the study

Any condition or situation, which, in the investigator's opinion, puts the patient at significant risk, could confound the study results, or may interfere significantly with the patient's participation in the study

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Degree of erectile dysfunction after surgery | up to one year
  Measured by changes in IIEF-5
Penile complications | up to one year
  Measured by questionnaire made for this study

SECONDARY OUTCOMES:
Occurrence of failure within the follow up period | One year
Occurrence of complications | From operation to one year

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Schultz, MD, Principal Investigator — Consultant
Locations (4):
- Helsinki University Hospital, Helsinki, Finland
- Oslo University Hospital, Dept of Urology, Oslo, Norway
- Sweden (2):
  - Sahlgrenska University Hospital, Dept of Urology, Gothenburg
  - Örebro University Hospital, Dept of Urology, Örebro